CLINICAL TRIAL: NCT03995316
Title: Responsive e-Health Intervention for Perinatal Depression in Healthcare Settings
Acronym: MMB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Behavioral Intervention Strategies, Inc. (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MH109191; 5R44MH109191-03 (NIH)
Record Dates: First submitted 2019-06-17; First posted 2019-06-24 (Actual); Results first posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Perinatal Depression
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: 2-Arm random control trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment As Usual + MMB 2.0 (Other): Women assigned to use MMB 2.0, along with NorthShore HealthSystem's well established usual care, will be guided by the program to move sequentially through 6 sessions, one of which becomes available for use each week, while interacting with engaging activities within each session along with recommended practice activities to encourage transfer of learning and skills to everyday routines. Content is presented using text, interactions, animations, and videos. MMB includes daily tracking and charting of mood and pleasant activities as well as online access to a library, covering a range of issues of concern to pregnant women and new mothers. Integrated text messages offer both motivational messages and links to access specific portions of session content in the MMB 2.0 program. The study coordinator will also provide up to 3 supportive coaching calls to each woman in the MMB 2.0 condition. These calls complement and thus are adjunctive to the MMB 2.0 program.
  Interventions: Behavioral: Treatment As Usual + MMB 2.0
- Treatment As Usual Only (Other): NorthShore HealthSystem's treatment as usual, or usual care, has been in place since 2003. Screen positive women randomized to this condition will receive social work assessment by phone, followed by community mental health referral as indicated. Referrals will vary by need and may include psychotherapy, support groups, or psychiatry. Referrals will include consideration of geographic proximity, insurance, and acuity. Consistent with routine practice, NorthShore staff will document time spent during evaluation and in making specific referrals.
  Interventions: Behavioral: Treatment As Usual Only

INTERVENTIONS:
Behavioral: Treatment As Usual + MMB 2.0 — Women assigned to use MMB 2.0, along with NorthShore HealthSystem's well established usual care, will be guided by the program to move sequentially through 6 sessions, one of which becomes available for use each week, while interacting with engaging activities within each session along with recommended practice activities to encourage transfer of learning and skills to everyday routines. Content is presented using text, interactions, animations, and videos. MMB includes daily tracking and charting of mood and pleasant activities as well as online access to a library, covering a range of issues of concern to pregnant women and new mothers. Integrated text messages offer both motivational messages and links to access specific portions of session content in the MMB 2.0 program. The study coordinator will also provide up to 3 supportive coaching calls to each woman in the MMB 2.0 condition. These calls complement and thus are adjunctive to the MMB 2.0 program.
  Arms: Treatment As Usual + MMB 2.0
Behavioral: Treatment As Usual Only — NorthShore HealthSystem's treatment as usual, or usual care, has been in place since 2003. Screen positive women randomized to this condition will receive social work assessment by phone, followed by community mental health referral as indicated. Referrals will vary by need and may include psychotherapy, support groups, or psychiatry. Referrals will include consideration of geographic proximity, insurance, and acuity. Consistent with routine practice, NorthShore staff will document time spent during evaluation and in making specific referrals.
  Arms: Treatment As Usual Only

SUMMARY:
Perinatal depression is experienced by at least 14-20% of pregnant and postpartum women, and is recognized as the most common complication of childbirth. In this project, the investigators plan to complete the process of making MomMoodBooster (MMB), a web-based cognitive-behavioral depression intervention, into a commercial ready product, MMB 2.0, that fits the workflow and staffing of healthcare organizations and is designed for both prenatal and postpartum women who are depressed. The investigators will also conduct a 2-arm randomized controlled trial to evaluate the efficacy of treatment as usual plus MMB 2.0 compared to treatment as usual in a large healthcare setting.

DETAILED DESCRIPTION:
Perinatal depression (experienced by at least 14-20% of pregnant and postpartum women) is recognized as the most common complication of childbirth and as having extremely serious consequences, including significant suffering for pregnant women/new mothers and their families, and adverse impacts on infant development. Unfortunately, there are many barriers that make it difficult for women with perinatal depression to access clinic-based mental health treatments, and participation is low. Treatment uptake is limited by psychological barriers (stigma, feelings of failure, and embarrassment); knowledge barriers (poor understanding about impact of perinatal depression on infant health, uncertainty about where to get treatment); infrastructure barriers (fear of negative judgment from care providers, avoidance of prescription medications while breastfeeding); physical barriers in rural settings (too few care providers, unacceptable logistical demands on time, transportation, and childcare); and provider-level barriers (inadequate skills, fear of liability, dearth of treatment options, and inadequate reimbursement). To address this need, investigators obtained funding (National Institutes of Health (NIH) R01MH084931) to develop and test the MomMoodBooster program (MMB), an innovative Web-based program for treating postpartum depression (PPD). Based on cognitive behavioral therapy (CBT) and incorporating multimedia modeling and engaging activities, MMB is designed to enable women to identify patterns in their thoughts and behaviors and to develop a personal action plan to make helpful changes. MMB also has an administrative website designed for use by both project managers and supportive phone coaches to monitor the overall progress of participants. In our Small Business Innovation Research (SBIR) Phase I grant (R43MH109191), the investigators began a redesign of MMB so that it could be used more effectively as a product for delivering PPD treatment by practical healthcare delivery organizations. Specifically, the investigators enhanced the underlying database architecture (and the related administration website interface) to make it easier for multiple organizations in multiple settings to use MMB. In our proposed SBIR Phase II, the investigators propose to complete the process of making a commercial-ready product (MMB 2.0) that fits the workflow and staffing of healthcare organizations. Specifically, the investigators propose to finish the enhancement of the database architecture and its administrative site, to expand MMB to include prenatal as well as postpartum depressed women, and to deliver MMB using a new responsive design technology so that women will be able to use it interchangeably with any internet-accessible computer device (desktop, laptop, tablet, smart-phone). Finally, the investigators plan to use a 2-arm randomized controlled trial to evaluate the efficacy of MMB 2.0 compared to treatment as usual in a large healthcare setting.

ELIGIBILITY:
Inclusion Criteria:

* pregnant or postpartum
* have elevated Edinburgh Postnatal Depression Scale (EPDS) of ≥ 12
* access to broadband internet and a computer at home (desktop, laptop, tablet) or a smartphone (iOS or Android)
* English language proficiency sufficient to enable completion of the informed consent and to engage in all study activities that are delivered in English

Exclusion Criteria:

* Women assessed with active suicidal ideation will be excluded and provided with immediate psychiatric care consistent with NorthShore's established safety protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - NorthShore University HealthSystem, Chicago, Illinois
  - Oregon Research Behavioral Intervention Strategies, Inc., Springfield, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Danaher BG, Seeley JR, Silver RK, Tyler MS, Kim JJ, La Porte LM, Cleveland E, Smith DR, Milgrom J, Gau JM. Trial of a patient-directed eHealth program to ameliorate perinatal depression: the MomMoodBooster2 practical effectiveness study. Am J Obstet Gynecol. 2023 Apr;228(4):453.e1-453.e10. doi: 10.1016/j.ajog.2022.09.027. Epub 2022 Sep 26. PMID 36174746

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment As Usual + MMB 2.0 | Treatment As Usual Only
Started | 96 | 95
Completed | 86 | 92
Not Completed | 10 | 3
Not completed — Lost to Follow-up | 10 | 3

BASELINE CHARACTERISTICS:
Population: The analyses population was intent-to-treat and thus does not differ from the randomized sample.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment As Usual + MMB 2.0 | Treatment As Usual Only | Total
Number analyzed (Participants) | 96 | 95 | 191
Age, Categorical [Count of Participants; unit: Participants]
  Age: <=18 years | 0 | 0 | 0
  Age: Between 18 and 65 years | 96 | 95 | 191
  Age: >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Age determined from date of birth and date of baseline assessment.
  years | 31.7 (5.2) | 32.1 (5.4) | 31.9 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 95 | 191
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 11 | 23
  Not Hispanic or Latino | 78 | 79 | 157
  Unknown or Not Reported | 6 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 10 | 17 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 7 | 15
  White | 66 | 60 | 126
  More than one race | 8 | 8 | 16
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 96 | 95 | 191

OUTCOME MEASURES:

1. Primary Outcome: Change in Primary Health Questionnaire (PHQ-9)
Description: The PHQ-9 measures self-reports of depressive symptoms within the prior 2 weeks and has been well-validated, shown high test-retest reliability, shown high internal consistency, and shown to be responsive to changes in treatment. Response options are on a 4-point scale (0 = not at all, 3 = nearly every day). The minimum overall score is 0 and the maximum overall score for the PHQ-9 is 27. Higher values represent more severe depression status.
Time Frame: Pretest (at enrollment) and posttest (3 months post enrollment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment As Usual + MMB 2.0 | Treatment As Usual Only
Number analyzed (Participants) | 96 | 95
score on a scale
  Pretest | 10.68 (4.96) | 10.24 (5.57)
  Posttest | 5.78 (4.42) | 7.48 (5.67)
Statistical Analysis 1: Comparison: Treatment As Usual + MMB 2.0 vs Treatment As Usual Only; Test type: Superiority; p = .003, t-test, 2 sided; Slope = -0.76, Standard Error of Mean 0.25 — The slope value reflects the mean difference between conditions in the linear slope from the pretest to posttest assessment

2. Secondary Outcome: Change in General Anxiety Disorder (GAD)
Description: The 7-item GAD measures generalized anxiety. Response options are on a 4-point scale (0 = did not apply to me, 3 = applied to me most of the time). A total sum score was computed. The minimum overall score is 0 and the maximum overall score is 21. Higher values represent more severe symptoms of generalized anxiety.
Time Frame: Pretest (at enrollment) and posttest (3 months post enrollment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment As Usual + MMB 2.0 | Treatment As Usual Only
Number analyzed (Participants) | 96 | 95
score on a scale
  Pretest | 5.23 (3.90) | 5.96 (4.43)
  Posttest | 2.81 (2.82) | 4.12 (3.83)
Statistical Analysis 1: Comparison: Treatment As Usual + MMB 2.0 vs Treatment As Usual Only; Test type: Superiority; p = .283, t-test, 2 sided; Slope = -0.18, Standard Error of Mean 0.17 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change in Stress
Description: The 7-item stress will measure generalized stress. Response options are on a 4-point response option (0 = did not apply to me, 3 = applied to me most of the time). A total sum score was computed. The minimum overall score is 0 and the maximum overall score is 21. Higher values represent more severe symptoms of generalized stress.
Time Frame: Pretest (at enrollment) and posttest (3 months post enrollment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment As Usual + MMB 2.0 | Treatment As Usual Only
Number analyzed (Participants) | 96 | 95
score on a scale
  Pretest | 9.61 (4.05) | 10.36 (4.53)
  Posttest | 5.79 (3.47) | 8.10 (4.65)
Statistical Analysis 1: Comparison: Treatment As Usual + MMB 2.0 vs Treatment As Usual Only; Test type: Superiority; p = .019, t-test, 2 sided; Slope = -0.51, Standard Error of Mean 0.22 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change in Behavioral Activation for Depression Scale (BADS)
Description: The 9-item BADS measures self-reports of activation, avoidance/rumination, work/school impairment, and social impairments. Response options are on a 7-point scale (0 = nota at all, 6 = completely) and a total sum score was computed. The minimum overall score is 0 and the maximum overall score is 54. Higher values represent more severe depression status related to behavioral activation.
Time Frame: Pretest (at enrollment) and posttest (3 months post enrollment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment As Usual + MMB 2.0 | Treatment As Usual Only
Number analyzed (Participants) | 96 | 95
score on a scale
  Pretest | 25.15 (7.99) | 24.46 (8.66)
  Posttest | 31.15 (8.41) | 29.37 (9.41)
Statistical Analysis 1: Comparison: Treatment As Usual + MMB 2.0 vs Treatment As Usual Only; Test type: Superiority; p = .440, t-test, 2 sided; Slope = 0.34, Standard Error of Mean 0.44 — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Change in Automatic Thoughts Questionnaire - Short Form (ATQ)
Description: The 8-item ATQ measures negative thoughts associated with depression. Response options are on a 4-point scale (0 = not at all, 3 = all the time) and a total mean score was computed and can range from 0 to 3. Higher values represent more severe depression status related to experiencing automatic thoughts.
Time Frame: Pretest (at enrollment) and posttest (3 months post enrollment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment As Usual + MMB 2.0 | Treatment As Usual Only
Number analyzed (Participants) | 96 | 95
score on a scale
  Pretest | 1.23 (0.65) | 1.24 (0.66)
  Posttest | 0.72 (0.57) | 0.90 (0.55)
Statistical Analysis 1: Comparison: Treatment As Usual + MMB 2.0 vs Treatment As Usual Only; Test type: Superiority; p = .055, t-test, 2 sided; Slope = -0.06, Standard Error of Mean 0.03 — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Change in Self-Efficacy
Description: The 8-item self-efficacy score measures confidence in one's ability to implement the skills taught in the program (e.g., how confident are you that you can increase your daily pleasant activities?). Response options are on 5-point scale (1 = not at all confident, , 5 = Very confident) and scores were averaged across the 8-items and can range from 1 to 5. A higher score indicates more self-efficacy to perform the tasks taught in the program.
Time Frame: Pretest (at enrollment) and posttest (3 months post enrollment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment As Usual + MMB 2.0 | Treatment As Usual Only
Number analyzed (Participants) | 96 | 95
score on a scale
  Pretest | 2.86 (0.74) | 2.77 (0.73)
  Posttest | 3.40 (0.79) | 3.05 (0.78)
Statistical Analysis 1: Comparison: Treatment As Usual + MMB 2.0 vs Treatment As Usual Only; Test type: Superiority; p = .041, t-test, 2 sided; Slope = 0.08, Standard Error of Mean 0.04 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from completion randomization through the final 12-week assessment period.
Arm/Group | Treatment As Usual + MMB 2.0 | Treatment As Usual Only
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/95
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/95
Other Adverse Events (participants affected / at risk) | 0/96 | 0/95

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT03995316/Prot_SAP_000.pdf
  • Informed Consent Form (2018-01-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT03995316/ICF_001.pdf